CLINICAL TRIAL: NCT04544046
Title: Randomized Trial of a Supportive Oncology Care at Home Intervention for Patients With Cancer Receiving Definitive Treatment
Brief Title: Supportive Oncology Care At Home RCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Medically Home (Unknown)
Responsible Party: Principal Investigator, Ryan Nipp, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-331
Record Dates: First submitted 2020-09-03; First posted 2020-09-10 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Pancreatic Cancer; GastroEsophageal Cancer; Rectal Cancer; Head and Neck Cancer; Lymphoma
Keywords: Pancreatic Cancer; GastroEsophageal Cancer; Rectal Cancer; Head and Neck Cancer; Lymphoma
MeSH Terms: conditions — Pancreatic Neoplasms; Rectal Neoplasms; Head and Neck Neoplasms; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): Participants assigned to the standard care arm will receive standard oncology care and attend regular clinic visits. Participants on the standard care arm will complete questionnaires from baseline up to 6 months following enrollment.
  Interventions: Other: Usual Care
- Supportive Oncology Care at Home (Experimental): The research study procedures include:
  * Remote monitoring of symptoms, vitals, and body weight
  * Questionnaires asking about demographic information (e.g. gender, ethnicity, income) and experience with cancer (e.g. quality of life, symptoms)
  * Data collection from medical record
  Interventions: Other: Supportive Oncology Care at Home

INTERVENTIONS:
Other: Supportive Oncology Care at Home — Remote monitoring of symptoms, vital signs, and body weight with home-based care to address any concerning issues identified.
  Arms: Supportive Oncology Care at Home
Other: Usual Care — Standard care arm will receive standard oncology care and attend regular clinic visits.
  Arms: Usual Care

SUMMARY:
This research study is evaluating a program that entails remote monitoring and home-based care for people with cancer who are receiving chemotherapy, radiotherapy, or chemoradiotherapy.

DETAILED DESCRIPTION:
Participants receiving treatment for cancer often require multiple care visits and may experience significant symptoms and side-effects related to the cancer and the cancer treatment.

This research study is evaluating if a program that involves remote monitoring and home-based care may improve the quality of life, ability to manage symptoms, and overall care of individuals during cancer treatment. Remote monitoring is broadly defined as a way of monitor outside of conventional clinical settings (e.g. in the home) that often utilizes technology to increase access to care.

Eligible participants will be randomized into one of two groups:

* Usual Care or
* Supportive Oncology Care at Home

It is expected that about 300 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible, patients must be: age 18 or older
* Receiving definitive treatment (i.e. neoadjuvant chemotherapy and/or chemoradiation with curative intent) for pancreatic, gastroesophageal, rectal, head and neck cancer, or lymphoma
* Within two weeks of starting treatment
* Planning to receive care at Massachusetts General Hospital (MGH)
* Verbally fluent in English
* Residing within 50 miles of Massachusetts General Hospital

Exclusion Criteria:

* Patients with uncontrolled psychiatric illness or impaired cognition interfering with their ability to understand study procedures and provide written or electronic informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-09-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants requiring a hospital admission or emergency department visit | baseline to 6 months
  Compare the difference between study arms using Fisher's exact tests, and logistic regression, adjusted for any potential confounders that are imbalanced between the two groups at baseline (e.g. age, gender).

SECONDARY OUTCOMES:
Proportion of days participants spend outside of the hospital during the study period | baseline to 6 months
  Linear regression or Poisson regression based on normality of the data adjusted for any potential confounders that are imbalanced between the two groups (e.g. age, gender).
Proportion of patients needing an urgent visit to clinic | baseline to 6 months
  Linear regression or Poisson regression based on normality of the data adjusted for any potential confounders that are imbalanced between the two groups (e.g. age, gender).
Rate of treatment delays | baseline to 6 months
  Compare rates of treatment interruptions (e.g. delays) using Fisher's exact tests and logistic regression, adjusted for any potential confounders that are imbalanced between the two groups at baseline (e.g. age, gender).
Comparison of dose intensity | baseline to 6 months
  Compare dose intensity using linear regression or Poisson regression based on normality of the data adjusted for any potential confounders that are imbalanced between the two groups (e.g. age, gender).
Change in symptom burden (ESAS) | baseline up to 6 months
  Linear regression or Poisson regression based on normality of the data adjusted for baseline values of each respective patient-reported outcome and any potential confounders that are imbalanced between the two groups (e.g. age, gender).
Change in quality of life (FACT-G) | baseline to 6 months
  Linear regression or Poisson regression based on normality of the data adjusted for baseline values of each respective patient-reported outcome and any potential confounders that are imbalanced between the two groups (e.g. age, gender).
Change in psychological distress (HADS) | baseline to 6 months
  Linear regression or Poisson regression based on normality of the data adjusted for baseline values of each respective patient-reported outcome and any potential confounders that are imbalanced between the two groups (e.g. age, gender).
Change in care satisfaction (FAMCARE) | baseline to 6 months
  Linear regression or Poisson regression based on normality of the data adjusted for baseline values of each respective patient-reported outcome and any potential confounders that are imbalanced between the two groups (e.g. age, gender).
Change in Activities of Daily Living (ADLs) | baseline to 6 months
  Linear regression or Poisson regression based on normality of the data adjusted for baseline values of each respective patient-reported outcome and any potential confounders that are imbalanced between the two groups (e.g. age, gender).
Change in Instrumental Activities of Daily Living (IADLs) | baseline to 6 months
  Linear regression or Poisson regression based on normality of the data adjusted for baseline values of each respective patient-reported outcome and any potential confounders that are imbalanced between the two groups (e.g. age, gender).

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Nipp, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: MGH - Contact the Partners Innovations team at http://www.partners.org/innovation

REFERENCES:
- [Derived] Nipp RD, Shulman E, Smith M, Brown PMC, Johnson PC, Gaufberg E, Vyas C, Qian CL, Neckermann I, Hornstein SB, Reynolds MJ, Greer J, Temel JS, El-Jawahri A. Supportive oncology care at home interventions: protocols for clinical trials to shift the paradigm of care for patients with cancer. BMC Cancer. 2022 Apr 9;22(1):383. doi: 10.1186/s12885-022-09461-z. PMID 35397575